CLINICAL TRIAL: NCT03573011
Title: PSMA-PET/CT for Prostate Cancer - Phase 2 Trial
Brief Title: PSMA PET/CT for Prostate Cancer
Acronym: NGP2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: AGO/2017/006 phase 2 trial; 2017-003461-96 (EudraCT Number)
Record Dates: First submitted 2018-06-19; First posted 2018-06-28 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-01

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; biochemical recurrence; 18F-PET imaging
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Original phase 2 (44 subjects) Concerning the dose of [18F]PSMA-11, half of the patients in the phase 2 study will be injected with 2.0 ± 0.2 MBq/kg bodyweight. The other half will be injected with 4.0 ± 0.4 MBq/kg body weight. Randomization of patients to one of these two groups will be performed using a block randomization design with block sizes of two, four, and six.
  Extension phase 2 (22 subjects):
  For this part of the phase 2 study, all patients will be injected with 2.0 ± 0.2 MBq/kg bodyweight [18F]PSMA-11. No Randomisation or masking is applicable for this group of 22 subjects.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Original phase 2 trial (44 subjects)
  The assigned [18F]PSMA-11 dosing group will be blind to the recruiting physicians, the patient the staff member(s) while planning the [18F]PSMA-11 scanday of the patient, and the nuclear medicine physicians interpreting the images.
  Next to the clinical trial coordinators, also the staff members responsible for the preparation of the individual [18F]PSMA-11 dose and the IV injection of this dose are aware of the dose group (2.0 ± 0.2 or 4.0 ± 0.4 MBq/kg body weight), which means that they are NOT blinded. However, these staff members do not carry out any further study specific handlings.
  Extension phase 2 trial (22 subjects):
  masking is not applicable for this part of the phase 2 trial.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2.0 ± 0.2 MBq/kg [18F]PSMA-11 dosing group (Experimental): To define the optimal [18F]PSMA-11 scan protocol, the quality of the PET images from patients that received 2.0 ± 0.2 MBq/kg will be compared to the images from patients that received 4.0 ± 0.4 MBq/kg.
  Patients in this study arm will receive 2.0 ± 0.2 MBq/kg for acquiring the [18F]PSMA-11 scan. All other study parameters and procedures are identical to those in the other study arm.
  As for the use of radiopharmaceuticals, the ALARA ('as low as reasonably achievable') principle must be applied, this study arm is considered to be the reference.
  Interventions: Diagnostic Test: [18F]PSMA-11
- 4.0 ± 0.4 MBq/kg [18F]PSMA-11 dosing group (Experimental): Concerning the dose of [18F]PSMA-11, the patients in this study arm will receive 4.0 ± 0.4 MBq/kg for the [18F]PSMA-11 scan. All other study parameters and procedures are identical to those in the other study arm
  Interventions: Diagnostic Test: [18F]PSMA-11

INTERVENTIONS:
Diagnostic Test: [18F]PSMA-11 — 18F-PET imaging

SUMMARY:
Prostate cancer is the most frequently occurring male cancer in Belgium. Patients who have been treated for prostate cancer, i.e. by surgery and/or radiotherapy, in a substantial degree suffer from a tumor recurrence, often diagnosed by an increase in serum tumor marker Prostate Specific Antigen (PSA) within the first few years. In these patients with evidence of a tumor recurrence after primary treatment, it is important to most exactly define the location(s) of tumor, to guide appropriate therapy by surgery, radiotherapy and/or hormonotherapy. In so-called oligo-metastatic disease targeted therapy may still be curative and prevent the disease from spreading to distant locations. Therefore it is of paramount importance to have an accurate tool of medical imaging to localize all possible locations to be treated.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with prostate cancer, either in the setting of diagnosis of biochemical recurrence after previous treatment, or at primary diagnosis and staging.

Exclusion Criteria:

* Age: <18 years
* Physically or mentally unfit to perform the sequential procedures
* Refusal of patient to be informed about accidental findings on scans
* Patients with heart failure if ejection fraction < 45% (phase 2 trial)
* History of anaphylactic shock after administration of Visipaque CT contrast (phase 2 trial)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — male with prostate cancer
Enrollment: 64 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2019-02-18 (Actual)

PRIMARY OUTCOMES:
Evaluation of effective targeting of prostate cancer and eventual metastases | 0 to 3.5 hours post radiotracer injection
  Two PET/CT scans with [18F]PSMA-11 will be acquired to evaluate the effectiveness of targeting prostate cancer and eventual metastases
Determination of the optimal scan protocol: define optimal time of scanning | 0 to 3.5 hours post radiotracer injection
  Based on the quality of the images and feasibility of tumor targetting (4 point '0-3' scoring scale - higher score represents a higher intensity lesion), the optimal time (60 min or 180 min post radiotracer injection) will be defined
Determination of the optimal scan protocol: define optimal scan duration | 0 to 3.5 hours post radiotracer injection
  Based on the quality of the images and feasibility of tumor targetting (4 point '0-3' scoring scale, higher score represents a higher intensity lesion), the optimal scan duration (1.5 minutes/bed position or 3.0 minutes/bed position) will be defined
Determination of the optimal scan protocol: define optimal dose | 0 to 3.5 hours post radiotracer injection
  Based on the overall image quality (7 point '1-7' scoring scale for image blurriness, higher score represents a higher quality image), the optimal dose of [18F]PSMA-11 (2.0 or 4.0 MBq/kg) will be defined
Determination of the optimal scan protocol: evaluation of the added value of furosemide (to improve diuresis), as part of the standard scanprotocol | 0 to 1.5 hours post radiotracer injection
  Based on the degree that the radiotracer uptake in the bladder and in the ureters is disruptive for the interpretation of the scan (visual interpretation by nuclearist using a 7 point '1-7' scoring scale, higher score equals a more pronounced disturbance), the added value of furosemide, as part of the standard scanprotocol, will be defined

SECONDARY OUTCOMES:
Evaluation of the inter-observer difference for interpretation of [18F]PSMA-11 scans | 0 - 60 days post [18F]PSMA-11 administration
  The inter-observer difference for analysing the [18F]PSMA-11 PET images will be investigated between at least two nuclear physicians. Results will be expressed as a cohen's kappa
Evaluation of the diagnostic specificity of [18F]PSMA-11 | 0 - 60 days post [18F]PSMA-11 administration
  Following the [18F]PSMA PET/CT scans in the phase 2 trial, the treating physician will continue the follow-up and treatment of the patient. Hereby, depending of the selected conventional treatment or procedure, the following data will be also collected (if available within 60 days following the day of the [18F]PSMA scan) to investigate the diagnostic specificity of [18F]PSMA-11:
  * In case the treating physician opts to perform a radical prostatectomy or lymphadenectomy or to take a biopt, the anatomopathological diagnosis (PSMA expression in tissue) will be used as an endpoint for correlation with the results of the [18F]PSMA scan.
  * In case the treating physician opts for radiotherapy or hormone therapy, the (change in) PSA levels will be used as an endpoint for correlation with the results of the [18F]PSMA scan.
  * In case the treating physician opts to acquire an additional MRI, suspicious lesions on the MRI will be also compared with those observed on the [18F]PSMA PET/CT scan.
Evaluation of the impact of the [18F]PSMA-11 scan on the choice of therapy | Pre [18F]PSMA-11 PET management plan: between the date the patient signed the informed consent form and the date of the [18F]PSMA-11 scan. Post [18F]PSMA-11 PET management plan: 0 - 60 days post [18F]PSMA-11 administration
  The treating physician must fill in a questionnaire concerning the patients 'pre [18F]PSMA-11 PET' management plan. After the scan, the physician must fill in a second part of the questionnaire concerning how the [18F]PSMA-11 scan would influence the patient's treatment plan.

CONTACTS AND LOCATIONS:
Overall Officials: Piet Ost, Prof., Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, East Flanders, Belgium

REFERENCES:
- [Derived] Piron S, De Man K, Schelfhout V, Van Laeken N, Kersemans K, Achten E, De Vos F, Ost P. Optimization of PET protocol and interrater reliability of 18F-PSMA-11 imaging of prostate cancer. EJNMMI Res. 2020 Feb 24;10(1):14. doi: 10.1186/s13550-020-0593-7. PMID 32095919